CLINICAL TRIAL: NCT06999902
Title: A Double-Blind, Randomized, Multicenter, Trial Evaluating the Efficacy and Safety of PRAX-628 in Adults With Focal Seizures (POWER1)
Brief Title: Double-blind, Randomized Trial of PRAX-628 in Adults With Focal Seizures to Evaluate Efficacy and Safety (POWER1)
Acronym: POWER1
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-628-321
Record Dates: First submitted 2025-03-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Focal Seizure
Keywords: Focal Seizure
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Randomized, Double-Blind 20mg/day for 6 weeks then 30mg/day for remaining 6 weeks PRAX-628 (Experimental): Participants who meet all eligibility criteria will be randomized at Visit 1 (Day 1) to receive 20 mg of PRAX-628 for 6 weeks followed by 30 mg PRAX 628 for the remaining 6 weeks.
  Interventions: Drug: 20mg/day PRAX-628 for 6 weeks then 30mg/day PRAX-628 for remaining 6 weeks
- Randomized, Double-Blind Placebo (Experimental): Participants who meet all eligibility criteria will be randomized at Visit 1 (Day 1) to receive a matching placebo throughout the 12-week Treatment Period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 20mg/day PRAX-628 for 6 weeks then 30mg/day PRAX-628 for remaining 6 weeks — Once daily oral
  Arms: Randomized, Double-Blind 20mg/day for 6 weeks then 30mg/day for remaining 6 weeks PRAX-628
Drug: Placebo — Once daily oral
  Arms: Randomized, Double-Blind Placebo

SUMMARY:
A Double-Blind, Randomized, Multicenter, Trial Evaluating the Efficacy and Safety of PRAX-628 in Adults With Focal Seizures (POWER1)

DETAILED DESCRIPTION:
PRAX-628-321 (POWER1) is a double-blind, randomized, multicenter, trial to evaluate the efficacy and safety of PRAX-628 in adults who can attest to concurrently taking at least 1, but no more than 3 acceptable anti-seizure medications.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of focal onset epilepsy according to the International League Against Epilepsy (ILAE) Classification of Epilepsy.
2. Past evidence by computed tomography (CT) or magnetic resonance imaging (MRI) that has ruled out a progressive cause of epilepsy in the judgement of the investigator and/or in consultation with the medical monitor.

Exclusion Criteria:

1. Subject has had any of the of the following within the 12-month period preceding trial entry: History of pseudo or psychogenic seizures, cluster seizures where the individual seizures cannot be counted, an episode of convulsive status epilepticus requiring hospitalization and intubation, or subject only has focal seizures with awareness that do not have motor activity.
2. Planned epilepsy surgery during the course of the clinical trial.
3. History of neurosurgery for seizures <1 year prior to enrollment, or radiosurgery <2 years prior to enrollment or vagus nerve stimulation (VNS) implantation.
4. History of schizophrenia, obsessive-compulsive disorder, or other serious mental health disorders.
5. History of malignancy, myeloproliferative or lymphoproliferative disorders within the past 5 years are excluded.
6. History of cardiac disease(s)/cardiac conduction disorders/or cardiac structural abnormality(ies).
7. Has a positive test result or a known history of a positive test result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV) antibody at Screening.
8. Is pregnant or is breastfeeding at the time of Screening or has a positive serum pregnancy test at Screening or is planning to become pregnant during the clinical trial or within 14 days of the last study drug dose.
9. Has received any other experimental or investigational drug, device or other therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening, or any prior use of gene therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of PRAX-628 compared to placebo on focal seizure frequency in adults currently taking 1 to 3 ASMs | 12 weeks
  Median percent change in monthly (28 days) focal seizure frequency from the Screening/Observation Period to the Treatment Period for PRAX-628 compared to placebo.

SECONDARY OUTCOMES:
To evaluate the efficacy of PRAX 628 compared to placebo on focal seizure frequency in adults currently taking 1 to 3 ASMs | 12 weeks
  Proportion of participants experiencing a ≥50% reduction in monthly (28 days) focal seizure frequency from the Screening/Observation Period to the Treatment Period (Responder Rate) for PRAX 628 compared to placebo.
To assess trends over time in efficacy of PRAX 628 on focal seizure frequency | 12 weeks
  Percent change in monthly focal seizure frequency from the Screening/Observation Period to the Treatment Period for PRAX-628 compared with placebo.
To evaluate the efficacy of PRAX 628 compared to placebo on focal seizure frequency in adults currently taking 1 to 3 ASMs | 12 weeks
  Number of days post-randomization to reach the same number of monthly focal seizures as the Screening/Observation Period through the end of the Treatment Period
  Proportion of participants experiencing seizure freedom, 100% reduction in monthly (28 days) focal seizure frequency from the Screening/Observation Period to the Treatment Period for PRAX-628 compared with placebo
  Impact of PRAX-628 compared to placebo on PGI-S and CGI-S
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Incidence and severity of TEAEs, including discontinuation of study drug due to TEAEs
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Change in tympanic temperature in Celsius
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Change in heart rate in beats per minute
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Change in blood pressure in mm/Hg
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Change in respiratory rate in breaths per minute
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  The principal investigator (PI) or sub investigator will review the laboratory report and document this review. Any clinically significant adverse changes occurring during the clinical trial will be documented as adverse events.
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Incidence of clinically significant ECG abnormalities
To assess the safety and tolerability of PRAX-628 in adults with focal seizures | 12 weeks
  Changes in suicidality, as assessed by C-SSRS

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Praxis Precision Medicines
Locations (22):
- United States (16):
  - Praxis Research Site, Phoenix, Arizona
  - Praxis Research Site, DeLand, Florida
  - Praxis Research Site, Miami Lakes, Florida
  - Praxis Research Site, Chicago, Illinois
  - Praxis Research Site, Lafayette, Louisiana
  - Praxis Research Site, Bethesda, Maryland
  - Praxis Research Site, Chesterfield, Missouri
  - Praxis Research Site, Ozark, Missouri
  - Praxis Research Site, Hackensack, New Jersey
  - Praxis Research Site, Middletown, New York
  - Praxis Research Site, Canton, Ohio
  - Praxis Research Site, Oklahoma City, Oklahoma
  - Praxis Research Site, El Paso, Texas
  - Praxis Research Site, Frisco, Texas
  - Praxis Research Site, Round Rock, Texas
  - Praxis Research Site, Seabrook, Texas
- Spain (6):
  - Praxis Research Site, Barcelona
  - Praxis Research Site, Granda
  - Praxis Research Site, Madrid
  - Praxis Research Site, Málaga
  - Praxis Research Site, Terrassa
  - Praxis Research Site, Valencia